CLINICAL TRIAL: NCT07101120
Title: A Phase 2, Two-Part (Open-Label Followed by Double-Blind) Study Evaluating the Safety, Tolerability, Pharmacokinetics, and Efficacy of KH607 in the Treatment of Adult Participants With Moderate or Severe Major Depressive Disorder
Brief Title: A Phase 2 Study to Evaluate Efficacy and Safety of KH607 Tablets in Adult Participents With Major Depressive Disorder
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Chengdu Kanghong Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KH607-40101
Record Dates: First submitted 2025-07-24; First posted 2025-08-03 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-08

CONDITIONS: Major Depressive Disorder (MDD)
MeSH Terms: conditions — Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Part A: KH607 (Experimental): Participants receive KH607, 30 milligrams (mg), oral tablets, once daily for 14 days, as tolerated.
  Interventions: Drug: KH607 tablets
- Part B: Placebo (Placebo Comparator): Eligible participants receive matching placebo tabels once daily for 21 days.
  Interventions: Drug: placebo
- Part B: KH607 30mg (Experimental): Participants receive KH607, 30 milligrams (mg), oral tablets, once daily for 21 days.
  Interventions: Drug: KH607 tablets
- Part B: KH607 20mg (Experimental): Participants receive KH607, 20 milligrams (mg), oral tablets, once daily for 21 days.
  Interventions: Drug: KH607 tablets

INTERVENTIONS:
Drug: KH607 tablets — oral 30mg , once daily for 14 days
  Arms: Part A: KH607
Drug: placebo — oral, once daily for 21 days
  Arms: Part B: Placebo
Drug: KH607 tablets — oral 20mg, once daily for 21 days
  Arms: Part B: KH607 20mg
Drug: KH607 tablets — oral 30mg, once daily for 21 days
  Arms: Part B: KH607 30mg

SUMMARY:
This is a two-part (open-label followed by double-blind) study evaluating the safety, tolerability, pharmacokinetics, and efficacy of KH607 in 120 participants diagnosed with moderate or severe Major Depressive Disorder.

DETAILED DESCRIPTION:
Part A is an open-label study with dosing of KH607 tablets for 14 days.

Part B is a randomized, double-blind, parallel-group, placebo-controlled study. Eligible participants will be randomized to KH607 group or placebo group for 21 days.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18 to 65 years old (inclusive), Male or female.
2. Participant with diagnosis of MDD as diagnosed by Structured Clinical Interview for Diagnostic and Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) , with symptoms that have been present for at least a 4-week period
3. Participant has a Hamilton Rating Scale for Depression (HAM-D) total score ≥24 at screening and Day 1 (prior to dosing).
4. Participants who is taking antidepressants must have stopped for 7 days or 5 half-lives of the antidepressant prior to Day 1.
5. Participant is willing to stop other antidepressant or antianxiety medications and any new pharmacotherapy regimens, including as-needed benzodiazepine anxiolytics and sleep aids, until after completion of the Day 42 visit.
6. Fully understand the procedures and sigh the informed consent.

key exclusion criteria：

1. Participant is currently at significant risk of suicide, or has attempted suicide associated with the current episode of MDD.
2. Participant has a history of treatment-resistant depression, defined as persistent depressive symptoms despite treatment with adequate doses of antidepressants from two different classes for an adequate amount of time.
3. Participant has active psychosis.
4. Participant had used modified electroconvulsive therapy (MECT), transcranial magnetic stimulation (TMS), vagus nerve stimulation (VNS), deep brain stimulation (DBS), light therapy, etc. within 1 month prior to Day 1.
5. Subject has a history of sleep apnea.
6. Participant has a medical history of bipolar disorder, schizophrenia, and/or schizoaffective disorder (such as olanzapine, risperidone, quetiapine, aripiprazole, eptifamol, ziprasidone, caliparazine, sodium valproate, lithium carbonate, etc.) within the current major depressive episode.
7. Participant has a clinically significant abnormal 12-lead ECG at the screening or baseline visits. NOTE: mean QT interval calculated using the Fridericia method (QTcF) of >450 msec in males or >470 msec in females will be the basis for exclusion from the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Change From Baseline in the 17-item Hamilton Rating Scale for Depression (HAM-D17) Total Score at Day 15 - Part A | Baseline to Day 15
  The HAM-D total score comprised a sum of 17 individual item scores.The total score could range from 0 to 52. Higher scores indicated a greater degree of depression. The analysis was performed in participants included in Part B of the study.
Change From Baseline in the 17-item Hamilton Rating Scale for Depression (HAM-D17) Total Score at Day 22 - Part B | Baseline to Day 22
  The HAM-D total score comprised a sum of 17 individual item scores.The total score could range from 0 to 52. Higher scores indicated a greater degree of depression. The analysis was performed in participants included in Part B of the study.

SECONDARY OUTCOMES:
Part A：Pharmacokinetic parameters of KH607 tablets (Cmax） | Part A: Day 1 to Day 21.
  Maximum observed plasma concentration following administration
Change From Baseline in the 17-item Hamilton Rating Scale for Depression (HAM-D17) Total Score at Day 15 - Part A | Part A: Day 15
  The HAM-D total score comprised a sum of 17 individual item scores.The total score could range from 0 to 52. Higher scores indicated a greater degree of depression. The analysis was performed in participants included in Part B of the study.
Change From Baseline in the 17-item Hamilton Rating Scale for Depression (HAM-D17) Total Score at all other time points - Part A | Part A: Day 3,8,12,21,28
  The HAM-D total score comprised a sum of 17 individual item scores.The total score could range from 0 to 52. Higher scores indicated a greater degree of depression. The analysis was performed in participants included in Part B of the study.
Change From Baseline in the Montgomery and Åsberg Depression Rating Scale (MADRS) Total Score at Day 15 and All Other Time Points - Part A | Part A: Day 3,8,12,15,21,28
  The MADRS was a ten-item diagnostic questionnaire which psychiatrists used to measure the severity of depressive episodes in participants with mood disorders. It was designed as an adjunct to the HAM-D, to be more sensitive than the Hamilton Scale to the changes brought on by antidepressants and other forms of treatment. Each item yielded a score of 0 to 6. The MADRS total score was calculated as the sum of the 10 individual item scores, which ranged from 0 to 60. Higher MADRS scores indicated more severe depression. A negative change from baseline indicated less severe depression. A positive change from baseline indicated more severe depression. The analysis was performed in participants included in Part A of the study.
Change From Baseline in Hamilton Anxiety Rating Scale (HAM-A) Total Score at All Time Points - Part A | Part A: Day 3,8,12,15,21,28
  The 14-item HAM-A was used to rate the severity of symptoms of anxiety. Each of the 14 items was defined by a series of symptoms, and measured both psychic anxiety (mental agitation and psychological distress) and somatic anxiety (physical complaints related to anxiety). Scoring for HAM-A was calculated by assigning scores of 0 (not present) to 4 (very severe), with a total score range of 0 to 56. The HAM-A total score was calculated as the sum of the 14 individual item scores. A negative change from baseline indicated less anxiety. A positive change from baseline indicated more anxiety. The analysis was performed in participants included in Part A of the study.
Percentage of Participants With Clinical Global Impression - Severity (CGI-S) Response - Part A | Part A: Day 3,8,12,15,21,28
  The CGI-S item employed a 7-point Likert scale to measure the overall severtity in the participant's condition. The analysis was performed in participants included in Part A of the study.
Percentage of Participants With Clinical Global Impression - Improvement (CGI-I) Response - Part A | Part A: Day 3,8,12,15,21,28
  The CGI-I item employed a 7-point Likert scale to measure the overall improvement in the participant's condition post-treatment. The investigator rated the participant's total improvement whether or not it was due entirely to drug treatment. The CGI-I was only rated at post-treatment assessments. By definition, all CGI-I assessments were evaluated against baseline conditions. CGI-I response was defined as having a CGI-I global improvement score of 1 (very much improved) or 2 (much improved). The analysis was performed in participants included in Part A of the study. Data is reported for participants who had CGI-I response.
Percentage of Participants With HAM-D Response - Part A | Part A: Day 3,8,12,15,21,28
  HAM-D response was defined as having a 50% or greater reduction from baseline in HAM-D total score. The analysis was performed in participants included in Part A of the study. Data is reported for participants who had HAM-D response.
Percentage of Participants With HAM-D Remission - Part A | Part A: Day 3,8,12,15,21,28
  HAM-D remission was defined as having a HAM-D total score of ≤7. The analysis was performed in participants included in Part A of the study.
Change From Baseline in the 17-item Hamilton Rating Scale for Depression (HAM-D17) Total Score at all other time points - Part B | Part B: Day 3,8,15,28,35,42
  The HAM-D total score comprised a sum of 17 individual item scores.The total score could range from 0 to 52. Higher scores indicated a greater degree of depression. The analysis was performed in participants included in Part B of the study.
Change From Baseline in the Montgomery and Åsberg Depression Rating Scale (MADRS) Total Score at Day 15 and All Other Time Points - Part B | Part B: Days3, 8, 15, 22,28,35 and 42
  The MADRS was a ten-item diagnostic questionnaire which psychiatrists used to measure the severity of depressive episodes in participants with mood disorders. It was designed as an adjunct to the HAM-D, to be more sensitive than the Hamilton Scale to the changes brought on by antidepressants and other forms of treatment. Each item yielded a score of 0 to 6. The MADRS total score was calculated as the sum of the 10 individual item scores, which ranged from 0 to 60. Higher MADRS scores indicated more severe depression. A negative change from baseline indicated less severe depression. A positive change from baseline indicated more severe depression. The analysis was performed in participants included in Part A of the study.
Change From Baseline in Hamilton Anxiety Rating Scale (HAM-A) Total Score at All Time Points - Part B | Part B: Days3, 8, 15, 22,28,35 and 42
  The 14-item HAM-A was used to rate the severity of symptoms of anxiety. Each of the 14 items was defined by a series of symptoms, and measured both psychic anxiety (mental agitation and psychological distress) and somatic anxiety (physical complaints related to anxiety). Scoring for HAM-A was calculated by assigning scores of 0 (not present) to 4 (very severe), with a total score range of 0 to 56. The HAM-A total score was calculated as the sum of the 14 individual item scores. A negative change from baseline indicated less anxiety. A positive change from baseline indicated more anxiety. The analysis was performed in participants included in Part A of the study.
Percentage of Participants With Clinical Global Impression - Severity (CGI-S) Response - Part B | Part B: Days3, 8, 15, 22,28,35 and 42
Percentage of Participants With Clinical Global Impression - Improvement (CGI-I) Response - Part B | Part B: Days3, 8, 15, 22,28,35 and 42
Percentage of Participants With HAM-D Response - Part B | Part B: Days3, 8, 15, 22,28,35 and 42
Percentage of Participants With HAM-D Remission - Part B | Part B: Days3, 8, 15, 22,28,35 and 42
Part A：Pharmacokinetic parameters of KH607 tablets（Tmax） | Part A: Day 1 to Day 21.
  Time to reach the maximum observed plasma concentration following administration
Part A：Pharmacokinetic parameters of KH607 tablets（AUC0-inf） | Part A: Day 1 to Day 21.
  The AUCs is the area under the plasma concentration-time curve from time 0 to the Infinity post-dose.

IPD SHARING:
Plan to Share IPD: Yes